CLINICAL TRIAL: NCT02468024
Title: JoLT-Ca A Randomized Phase III Study of Sublobar Resection (SR) Versus Stereotactic Ablative Radiotherapy (SAbR) in High Risk Patients With Stage I Non-Small Cell Lung Cancer (NSCLC), The STABLE-MATES Trial
Brief Title: JoLT-Ca Sublobar Resection (SR) Versus Stereotactic Ablative Radiotherapy (SAbR) for Lung Cancer
Acronym: STABLE-MATES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Timmerman, MD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 022015-069
Record Dates: First submitted 2015-06-01; First posted 2015-06-10 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pulmonary Surgical Procedures; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Surgery versus SAbR
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 lung surgery (Active Comparator): Sublobar Resection (SR)
  Interventions: Procedure: Lung Surgery
- Arm 2 radiation therapy (Experimental): Stereotactic Ablative Radiotherapy (SAbR)
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Procedure: Lung Surgery — Sublobar Lung Resection
  Other Names: SR
  Arms: Arm 1 lung surgery
Radiation: Radiation therapy — Stereotactic Ablative Radiotherapy, 54 Gy in 3 fractions
  Other Names: SAbR
  Arms: Arm 2 radiation therapy

SUMMARY:
To Determine if SAbR improves survival over SR in High Risk Operable Stage I NSCLC

DETAILED DESCRIPTION:
Stereotactic Ablative Radiotherapy has been shown in single institution phase II and matched cohort studies to be effective at controlling primary early lung cancer. Recent pooled analysis of both the STARS and ROSEL randomized trials comparing SABR versus lobectomy have shown a significantly improved 3-year survival with SABR, giving further impetus for successful completion of a randomized trial .

Pre-randomized trial- Patients will be screened and pre-randomized to either SR or SAbR. Informed consent will be obtained after patients are made aware of the randomized assignment. Despite pre-randomization prior to consent, patients maintain their right to accept or decline any/all study activities. Only consenting patients will be allowed to participate in study activities, including observation after either randomized treatments or observation after standard of care treatment, while those declining consent will be managed by their physician(s) off study.Patients will be accrued and followed for a minimum of 2-years after treatment.

ELIGIBILITY:
1.0 Inclusion Criteria

1.1 Age > 18 years.

1.2 ECOG/Zubrod performance status (PS) 0, 1, or 2 (reference Appendix C).

1.3 Radiographic findings consistent with non-small cell lung cancer, including lesions with ground glass opacities with a solid component of 50% or greater.

1.4 The primary tumor in the lung must be biopsy confirmed non-small cell lung cancer within 180 days prior to randomization.

1.5 Tumor ≤ 4 cm maximum diameter, including clinical stage IA and selected IB by PET or PET integrated with a simultaneous CT scan (PET-CT) of the chest and upper abdomen performed within 180 days prior to randomization (reference Appendix A & B). Repeat imaging within 90 days prior to randomization is recommended for re-staging but is not required based on institutional norms.

1.6 All clinically suspicious mediastinal N1, N2, or N3 lymph nodes (> 1 cm short-axis dimension on CT scan and/or positive on PET scan) confirmed negative for involvement with NSCLC by one of the following methods: mediastinoscopy, anterior mediastinotomy, EUS/EBUS guided needle aspiration, CT-guided, video-assisted thoracoscopic or open lymph node biopsy within 180 days of randomization.

1.7 Tumor verified by a thoracic surgeon to be in a location that will permit sublobar resection.

1.8 Tumor located peripherally within the lung. NOTE: Peripheral is defined as not touching any surface within 2 cm of the proximal bronchial tree in all directions. See bronchial tree diagram below. Patients with non-peripheral (central) tumors are NOT eligible.

1.9 No evidence of distant metastases.

1.10 Availability of pulmonary function tests (PFTs - spirometry, DLCO, +/- arterial blood gases) within 180 days prior to registration. Patients with tracheotomy, etc, who are physically unable to perform PFTs (and therefore cannot be tested for the Major criteria in 3.1.11 below) are potentially still eligible if a study credentialed thoracic surgeon documents that the patient's health characteristics would otherwise have been acceptable for eligibility as a high risk but nonetheless operable patient (in particular be eligible for sublobar resection).

1.11 To define eligibility of patients being at high risk for surgery, certain criteria must be met.

Any one (1) of the following major criteria will define the high risk status for eligibility:

Major Criteria

* FEV1 ≤ 50% predicted (pre-bronchodilator value)
* DLCO ≤ 50% predicted (pre-bronchodilator value)
* Study credentialed thoracic surgeon believes the patient is potentially operable but that a lobectomy or pneumonectomy would be poorly tolerated by the patient for tangible or intangible reasons. The belief must be declared and documented in the medical record prior to randomization.

If any of the major criteria are met, the patient is eligible based on high risk for surgery and minor criteria do not need to be considered. However, if no major criteria is met, at least two (2) minor criteria being met will also define eligibility for meeting the high risk status.

Any two (2) of the following minor criteria will define the high risk status for eligibility:

* Minor Criteria
* Age ≥75
* FEV1 51-60% predicted (pre-bronchodilator value)
* DLCO 51-60% predicted (pre-bronchodilator value)
* Pulmonary hypertension (defined as a pulmonary artery systolic pressure greater than 40mm Hg) as estimated by echocardiography or right heart catheterization
* Poor left ventricular function (defined as an ejection fraction of 40% or less)
* Resting or Exercise Arterial pO2 ≤ 55 mm Hg or SpO2 ≤ 88%
* pCO2 > 45 mm Hg
* Modified Medical Research Council (MMRC) Dyspnea Scale ≥ 3.

1.12 No prior intra-thoracic radiation therapy for previously identified intra-thoracic primary tumor (e.g. previous lung cancer) on the ipsilateral side. NOTE: Previous radiotherapy as part of treatment for head and neck, breast, or other non-thoracic cancer is permitted to the ipsilateral side so long as possible radiation fields would not overlap. NOTE: Radiotherapy to the contralateral lung is allowed so long as it was completed more than 3 years prior to randomization and there is no overlap of radiation fields.

1.13 Previous chemotherapy, radiotherapy, or surgical resection specifically for the lung cancer being treated on this protocol is NOT permitted.

1.14 No prior lung resection on the ipsilateral side.

1.15 Non-pregnant and non-lactating. Women of child-bearing potential must have a negative urine or serum pregnancy test prior to registration. Peri-menopausal women must be amenorrheic > 12 months prior to registration to be considered not of childbearing potential.

1.16 No prior invasive malignancy, unless disease-free for ≥ 3 years prior to registration (exceptions: non-melanoma skin cancer, in-situ cancers).

1.17 Ability to understand and sign a written informed consent.

2.0 Exclusion Criteria

2.1 Age <18

2.2 ECOG/Zubrod performance status (PS) greater than 3.

2.3 Radiographic findings with ground glass opacities and less than 50% solid component will be excluded.

2.4 The primary tumor in the lung, biopsy confirmed non-small cell lung cancer greater than 180 days prior to randomization.

2.5 Tumor > 5 cm maximum diameter, including clinical stage IA and selected IB by PET or PET integrated with a simultaneous CT scan (PET-CT) of the chest and upper abdomen and/or performed greater than 180 days prior to randomization.

2.6 Lymph node biopsy greater than 180 days prior to randomization.

2.7 Thoracic surgeon confirms unable to remove tumor with sublobar resection.

2.8 Tumor located non-peripheral (central) region of lung (see bronchial tree diagram in 3.1.8).

2.9 Evidence of distant metastases.

2.10 Pulmonary function test (PFT - spirometry, DLCO, +/- arterial blood gases) greater than 180 days prior to registration. Patients physically unable to perform PFT's, such as patients with tracheotomy, that do not have written documentation from study credentialed thoracic surgeon stating eligibility.

2.11 Patients that do not meet either Major criteria or Minor criteria.

2.12 Prior intra-thoracic radiation therapy on ipsilateral side. Radiotherapy to the contralateral lung completed less than 3 years prior to randomization, with radiation field overlap.

2.13 Prior chemotherapy, radiotherapy, or surgical resection specifically for the lung cancer being treated on this protocol.

2.14 Prior lung resection on the ipsilateral side.

2.15 Pregnant and lactating women.

2.16 Prior invasive malignancy and less than 3 years disease free prior to registration (unless non-melanoma skin cancer, in-situ cancers).

2.17 Unable to understand and/ or sign a written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years
  To test the hypothesis that the 3-year overall survival in high risk operable patients with Stage I NSCLC is greater in patient who undergo SAbR as compared to standard sublobar resection (SR).

SECONDARY OUTCOMES:
progression free survival | 5 years
  survival at 5-years for Stage I NSCLC who undergo SR or SAbR.
toxicity as assessed toxicity using the Common Toxicity Criteria | 3 years
  toxicity using the Common Toxicity Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Robert Timmerman, MD, Principal Investigator — UTSW Medical Center
Locations (50):
- United States (40):
  - UCSD, La Jolla, California
  - University of Colorado/Memorial, Aurora, Colorado
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Curtis and Elizabeth Anderson Cancer, Savannah, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Health Care, Lexington, Kentucky
  - University of Louisville Physicians, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Luminis Health Research Institute, Annapolis, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Beaumont, Royal Oak, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Meridian Health System, Neptune City, New Jersey
  - New York University Langone Medical Center, New York, New York
  - SUNY - Upsate Medical Centre, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western (University Hospitals Case Medical Center), Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Providence Health & Services/Oregon Clinic, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny, Pittsburgh, Pennsylvania
  - UPMC Health System, Pittsburgh, Pennsylvania
  - Mount Nittany, State College, Pennsylvania
  - Lifespan Oncology Clinical Research, Providence, Rhode Island
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Clement Zablocki VA Medical Center, Milwaukee, Wisconsin
- Australia (3):
  - St. Vincent's Hospital Melbourne, Fitzroy, Melbourne
  - St. Vincent's/Peter Mac, Fitzroy, Victoria
  - Barwon Health - Uni Hospital Geelong, Geelong, Victoria
- Canada (6):
  - Trillium Health Partners, Mississauga, Canada
  - Sunnybrook Health Sciences Centre, Toronto, Canada
  - Ottawa Hospital Cancer Center, Ottawa, Ontario
  - UHN-Toronto, Toronto, Ontario
  - Lawson Health Science Center, London, Ontario, Canada
  - CHUM, Montreal, Quebec
- The James Cook University Hospital, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elbanna M, Shiue K, Edwards D, Cerra-Franco A, Agrawal N, Hinton J, Mereniuk T, Huang C, Ryan JL, Smith J, Aaron VD, Burney H, Zang Y, Holmes J, Langer M, Zellars R, Lautenschlaeger T. Impact of Lung Parenchymal-Only Failure on Overall Survival in Early-Stage Lung Cancer Patients Treated With Stereotactic Ablative Radiotherapy. Clin Lung Cancer. 2021 May;22(3):e342-e359. doi: 10.1016/j.cllc.2020.05.024. Epub 2020 Jun 2. PMID 32736936